CLINICAL TRIAL: NCT06316284
Title: The Role of miRNAs in the Regulation of Oxidative Stress and Microvascular Reactivity in Chronic Kidney Disease
Brief Title: miRNA in Chronic Kidney Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Collaborators: University Hospital Center Osijek (Unknown)
Responsible Party: Principal Investigator, Ines Drenjancevic, Vice Dean for Science Faculty of Medicine Osijek, Josip Juraj Strossmayer University of Osijek
Other Study IDs: miRNA-CKD
Record Dates: First submitted 2024-03-02; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney diseases; miRNA; oxidative stress; hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, peripheral blood mononuclear cells (PBMCs)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic kidney disease group: Patients with stage 3-5 CKD (eGFR CKD-EPI <60 mL/min/1.73 m2)
- Healthy controls: Healthy normotensive patients (eGFR CKD-EPI >90 mL/min/1.73 m2, BP <140/90 mmHg)
- Hypertensive Group: Hypertensive patients without CKD (eGFR CKD-EPI >90 mL/min/1.73 m2, BP >140/90 mmHg)

SUMMARY:
Oxidative stress and endoplasmic reticulum (ER) stress play a key role in tubular damage in both acute kidney injury and chronic kidney disease (CKD). Oxidative stress in the kidneys promotes renal vascular remodeling and increases preglomerular resistance. These are key elements in hypertension, acute and chronic kidney injury, as well as diabetic nephropathy. Chronic renal hypoxia is highlighted as the final common pathway to end-stage renal disease (ESRD). MicroRNA molecules (miRNA) also play an important role in these processes. MicroRNAs (miRNAs) are regulators of gene expression and play a role in the progression of renal ischemia-reperfusion injury. Although the pathophysiological contribution of microRNAs (miRNAs) to kidney damage has also been highlighted, the effect of miRNAs on kidney damage under conditions of oxidative and ER stress remains understudied.

ELIGIBILITY:
Inclusion Criteria:

* healthy normotensive adults (eGFR CKD-EPI >90 mL/min/1.73 m2, BP <140/90 mmHg)
* hypertensive adults (eGFR CKD-EPI >90 mL/min/1.73 m2, BP >140/90 mmHg)
* patients with chronic kidney disease stage 3-5 (eGFR CKD-EPI< 60 mL/min/1.73 m2)

Exclusion Criteria:

* cardiovascular diseases, but hypertension
* diabetes
* cerebrovascular diseases
* peripheral artery disease

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with CKD and healthy controls, i.e. patients with hypertension without kidney damage (eGFR CKD-EPI > 90 mL/min/1.73 m2). Subjects and controls will be age- and gender-matched. Inclusion criteria for patients with CKD: the study will include patients having chronic kidney disease of the 3rd - 5th degree (eGFR CKD-EPI< 60 mL/min/1.73 m2).
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Systemic microvascular function | Day 1
  Skin microvascular reactivity assessed by Laser Doppler flowmetry (post-occlusive reactive hyperemia, iontophoresis of acetylcholine and sodium nitroprusside) - measured in perfusion units (PU)
Serum level of antixidant enzymesprotein concentration of SOD, CAT and glutathione-peroxidase | Day 1
  Serum protein concentration of superoxide disimutase (SOD), catalase (CAT) and glutathione-peroxidase (GPx).
Detecton of miRNA of interest | Day 1
  The database for miRNA will be searched, and the miRNA of interest will be selected, determined and detected.

SECONDARY OUTCOMES:
Body fluid compartments | at one time point
  Total body water (L), extracellular water (L), intracellular water (L) and plasma fluid volume (L) will be assessed using non-invasive bioimpedance analysis (BIA).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No